CLINICAL TRIAL: NCT00276523
Title: A Randomized Phase II Study of SCH 54031 in Surgically Resectable Squamous Cell Tumors of the Head and Neck
Brief Title: PEG-interferon Alfa-2b in Treating Patients With Stage II, Stage III, or Stage IV Head and Neck Cancer That Can Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CDR0000441020; MDA-ID-01450; ID01-450 (Other: MD Anderson Cancer Center); NCT00078416 (obsolete NCT alias)
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Head and Neck Cancer
Keywords: stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — peginterferon alfa-2b; Neoadjuvant Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (Active Comparator): Control (no treatment), conventional surgery.
  Interventions: Procedure: Conventional surgery; Procedure: Neoadjuvant therapy
- PEG-Intron 0.5 mg/kg (Experimental): PEG-interferon alfa-2b 0.5 mg/kg subcutaneously (SQ) once a week for 3 weeks, plus surgery.
  Interventions: Biological: PEG-interferon alfa-2b; Procedure: Conventional surgery; Procedure: Neoadjuvant therapy
- PEG-Intron 2.5 mg/kg (Experimental): PEG-interferon alfa-2b 2.5 mg/kg SQ once a week for 3 weeks, plus surgery.
  Interventions: Biological: PEG-interferon alfa-2b; Procedure: Conventional surgery; Procedure: Neoadjuvant therapy
- PEG-Intron 5.0 mg/kg (Experimental): PEG-interferon Alfa-2b 5 mg/kg SQ once a week for 3 weeks, plus surgery.
  Interventions: Biological: PEG-interferon alfa-2b; Procedure: Conventional surgery; Procedure: Neoadjuvant therapy

INTERVENTIONS:
Biological: PEG-interferon alfa-2b — Study medication begins on Day 1 and taken subcutaneously once each week with the last dose being taken within 1 week prior to surgery or biopsy.
  Other Names: SCH 54031
  Arms: PEG-Intron 0.5 mg/kg; PEG-Intron 2.5 mg/kg; PEG-Intron 5.0 mg/kg
Procedure: Conventional surgery — Participants on the control arm may undergo surgery at anytime within 3 weeks of randomization, and those randomized to PEG-Intron will undergo surgery on Days 16-22 following initiation of treatment.
Procedure: Neoadjuvant therapy

SUMMARY:
RATIONALE: SCH 54031 (PEG-interferon alfa-2b) may interfere with the growth of tumor cells and slow the growth of head and neck cancer. It may also stop the growth of head and neck cancer by blocking blood flow to the tumor. Giving PEG-interferon alfa-2b before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This randomized phase II trial is studying how well different doses of PEG-interferon alfa-2b work in treating patients with stage II, stage III, or stage IV head and neck cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the antiangiogenic effects of PEG-interferon alfa-2b, in terms of pre- and post-treatment levels of microvessel density (MVD), endothelial cell apoptosis, vascular endothelial growth factor (VEGF), interleukin-8, basic fibroblast growth factor (bFGF), Nuclear Factor-KappaB (NF-KB), matrix metalloproteinase/MMP-9, and NF-KB in biopsy specimens, from patients with resectable stage II-IV squamous cell carcinoma of the head and neck.

Secondary

* Determine the toxicity profile of this drug in these patients.
* Determine the clinical response in patients treated with this drug.

OUTLINE: This is a randomized, controlled study. Patients are randomized to 1 of 4 treatment arms.

* Arm I: Patients undergo surgery within 3 weeks after randomization.
* Arm II: Patients receive PEG-interferon alfa-2b subcutaneously on days 1, 8, and 15.
* Arm III: Patients receive PEG-interferon alfa-2b as in arm II but at a higher dose.
* Arm IV: Patients receive PEG-interferon alfa-2b as in arm II but at a higher dose than in arm III.

In arms II, III, and IV, patients undergo surgery within 1 week after completion of PEG-interferon alfa-2b.

After completion of study treatment, patients are followed for up to 30 days.

PROJECTED ACCRUAL: A maximum of 72 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the head and neck

  * Stage II, III, or IV disease
  * One of the following primary tumor sites:

    * Oral cavity
    * Oropharynx
    * Hypopharynx
    * Larynx
* Resectable disease

  * Scheduled to undergo surgery as primary treatment

    * Distant metastases or a second primary tumor allowed provided tumor deemed resectable by the surgeon
* No squamous cell carcinoma of the nasopharynx or skin

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* White Blood Cells (WBC) > 3,000/mm^3
* Platelet count ≥ 150,000/mm^3
* Hemoglobin ≥ 10 g/dL

  * Transfusion and/or epoetin alfa support allowed provided it is given ≥ 1 week before study entry AND the patient is stable
* Bilirubin < 1.5 times upper limit of normal (ULN)
* serum glutamic pyruvic transaminase (SGPT) ≤ 5 times ULN
* Creatinine < 1.5 times ULN
* No hemolytic anemia
* No hemoglobinopathies (e.g., thalassemia)
* No prior or current ascites
* No bleeding varices
* No other evidence of decompensated liver disease
* No symptomatic ischemic heart disease
* No symptomatic congestive heart failure
* No other uncontrolled heart condition
* No chronic obstructive pulmonary disease
* No documented pulmonary hypertension
* No other chronic pulmonary disease
* No known HIV positivity
* No AIDS-related illness
* No active uncontrolled infection
* No immunologically mediated disease, including any of the following:

  * Inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis)
  * Rheumatoid arthritis
  * Idiopathic thrombocytopenia purpura
  * Systemic lupus erythematosus
  * Autoimmune hemolytic anemia
  * Scleroderma
  * Severe psoriasis
* No Central Nervous System (CNS) trauma
* No confusion or disorientation
* No active seizure disorders requiring medication
* No spontaneous encephalopathy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No pre-existing uncontrolled thyroid abnormality
* No poorly controlled diabetes mellitus
* No history of major psychiatric illness that would prelude giving informed consent
* No nonmalignant systemic disease that would preclude study participation

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior biologic therapy and recovered
* More than 4 weeks since prior chemotherapy and recovered
* More than 4 weeks since prior radiotherapy and recovered
* More than 4 weeks since prior surgery
* No prior interferon
* No other concurrent immunotherapy
* No concurrent chemotherapy
* No concurrent hormonal antineoplastic therapy
* No concurrent systemic corticosteroids
* No concurrent radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2004-02; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Response rate | 3 weeks following treatment

SECONDARY OUTCOMES:
Toxicity | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Roy S. Herbst, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M.D. Anderson Cancer Center at University of Texas, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Official Website — http://www.mdanderson.org